CLINICAL TRIAL: NCT06246799
Title: Comparative Effectiveness of Two Initial Combination Therapies in Patients With New Onset Diabetes
Brief Title: Comparative Effectiveness of Two Initial Combination Therapies in Patients With Recent Onset Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00000139; R01DK097554 (NIH)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes (Adult Onset)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; Pioglitazone; Sitagliptin Phosphate

STUDY DESIGN:
Intervention Model Description: Randomized open label study. There are 2 groups, with 2 sub groups, 1A, 1B and 1C included within Group 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group IC (Experimental): Tirzepatide starting at 2.5mg weekly titrated to 15mg weekly (2.5 month 1, 5mg month 2, 10mg month 3 and 15mg at month 4) with Pioglitazone beginning at 15mg daily and ending at 45mg daily (15mg month 1, 30mg month 2 and 45mg at month 3 onwards).
  Interventions: Drug: Tirzepatide; Drug: Pioglitazone
- Group II (Active Comparator): Metformin starting at 1000mg XR daily and Sitagliptin 100mg daily at week 4, Metformin will be increased to 200mg.
  Interventions: Drug: Sitagliptin; Drug: Metformin HCI XR
- Group IA (Active Comparator): Tirzepatide will be started at 2.5mg and increased to 15mg by month 4. At month 6, Pioglitazone will be added to the Tirzepatide, 15 mg daily.
  Interventions: Drug: Tirzepatide; Drug: Pioglitazone
- Group 1B (Active Comparator): Pioglitazone will be started at 15mg and increased to 45 mg by month 3. At month 6, tirzepatide 2.5mg will be started and increased weekly as tolerated.
  Interventions: Drug: Tirzepatide; Drug: Pioglitazone

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide:Participants will be initiated on 2.5mg weekly and increase their dose to 5mg at week 4, 10mg at week 8 and 15mg at week 12 as tolerated.
  Other Names: Mounjaro
  Arms: Group 1B; Group IA; Group IC
Drug: Pioglitazone — Pioglitazone: Participants will begin therapy at 15mg daily for the first 4 weeks then increase dose to 30mg at week 4 and to 45 mg at week 8, as tolerated.
  Other Names: Actos
  Arms: Group 1B; Group IA; Group IC
Drug: Sitagliptin — Sitagliptin: will be administered as a 100mg dose once daily.
  Other Names: Januvia
  Arms: Group II
Drug: Metformin HCI XR — Metformin will be administered at a dose of 1000mg for the first 4 weeks and then the dose increased to 2000mg.
  Other Names: Extended Release Metformin
  Arms: Group II

SUMMARY:
The primary purpose of this study is to evaluate the efficacy, durability, and mechanism of HbA1c reduction produced by the combination of pioglitazone plus tirzepatide compared to metformin plus sitagliptin in patients with recently diagnosed type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized open label controlled 2 arm study (with one of the arms containing 3 sub-groups) which aims to examine the effectiveness and long term effects on HbA1c reduction produced by the combination of pioglitazone plus tirzepatide versus metformin plus sitagliptin in recently diagnosed type 2 diabetes mellitus (T2DM) patients.

A subgroup of patients from group 1 will be invited to participate in a sub-study which lasts for 6 months and aims at exploring the metabolic/molecular mechanisms responsible for the study results. The selection of subjects to each subgroup will be done randomly and the end of sub-study, subjects will continue therapy and follow-up from month 6 on in the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Males and females; Age 18-75 years
3. Recently (within 5 years) diagnosed Type 2 Diabetes Mellitus (T2DM) patients
4. Drug naïve or receiving metformin monotherapy
5. HbA1c >6.5% (no limit on upper HbA1c value);
6. Willingness to adhere to the investigational product regimen
7. Good general health
8. Stable body weight over the preceding 3 months
9. Agreement to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

1. positive anti-GAD (antibodies to glutamic acid decarboxylase)
2. pregnancy or plan of becoming pregnant
3. evidence of proliferative diabetic retinopathy,
4. plasma creatinine >1.4 females or >1.5 males;
5. presence of congestive heart failure (CHF);
6. history of cancer (<5 years);
7. prior history of pancreatitis,
8. bladder cancer or family history of thyroid tumors;
9. presence of hematuria in the urine analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
number of subjects achieving HbA1c <6.5% at 6 months (Efficacy) | 6 months
  Therapy failure will be determined as HbA1c >6.5% in two consecutive HbA1c measurements 3 months apart. Time to cumulative incidence of therapy failure curves will be created in subjects receiving pioglitazone/tirzepatide versus subjects receiving metformin/sitagliptin
Number of subjects failing to achieving HbA1c <6.5% Long-term | month 60
  The failure to achieving HbA1c <6.5% (Durability) at the end of study in subjects receiving pioglitazone/tirzepatide (Group I) versus metformin/sitagliptin (Group II) in two consecutive HbA1c measurements 3 months apart.

SECONDARY OUTCOMES:
Change in insulin sensitivity | from baseline to end of study (60 months)
  Matsuda Index of insulin sensitivity or total glucose disposal measured with the clamp.These are the gold standard methods for quantification insulin sensitivity with the OGTT or a euglycemic clamp
Change in Beta Cell Function | Baseline to end of study (60 months)
  A calculated value using plasma glucose, insulin and C-peptide concentrations during the Oral Glucose Tolerance Test (OGTT) test.
Change in body weight | Baseline to end of study (60 months)
  Change from study beginning to end, measured in kilograms (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Abdul-Ghani, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - University Health System Texas Diabetic Institute, San Antonio, Texas
  - UT Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers at study completion when all data are analyzed and as summary results in ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP
Time Frame: At study completion at the time of publication.